CLINICAL TRIAL: NCT01547689
Title: Open-Label, Single-Center, Self Control, Phase Ⅰ/Ⅱ Clinical Trial to Evaluate the Safety and the Efficacy of UC-MSC in Patients With Alzheimer's Disease
Brief Title: Safety and Efficiency of Umbilical Cord-derived Mesenchymal Stem Cells(UC-MSC) in Patients With Alzheimer's Disease
Acronym: SEMAD
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Collaborators: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 307-CTC-MSC-001; 2011AA020114 (Other Grant/Funding Number: The "863 Projects" of MOST of PR China)
Record Dates: First submitted 2012-03-05; First posted 2012-03-08 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Human Umbilical Cord Derived MSC (Experimental)
  Interventions: Biological: Human Umbilical Cord Derived MSC

INTERVENTIONS:
Biological: Human Umbilical Cord Derived MSC — 20 million cells per subject（0.5×10^6 UC-MSCs per kg ） intravenous injection Infusion number:8 (Once every two weeks in the first month of each quarter) Time interval: two and a half months
  Other Names: Other Name: UC-MSC

SUMMARY:
The primary purpose of this study is to evaluate the safety and the tolerability of UC-MSC (Human Umbilical Cord-Derived Mesenchymal Stem Cell) .This study is also to investigate the efficacy of this treatment in patients with Alzheimer's disease (AD).

DETAILED DESCRIPTION:
To date, most AD patients who seek treatment already have neuritic plaques, neurofibrillary tangles, and neurodegeneration. At this stage of the disease, perhaps a multi-faceted approach to halt the toxicity of amyloid-β peptides and promote cell survival and/or replace lost cells would be most beneficial.Most of the treatments for Alzheimer disease are chemical drug which can improve the symptoms but is not able to inhibit the disease progression.

Mesenchymal stem cells (MSCs) are multipotent cells that are being clinically explored as a new therapeutic for treating a variety of immune-mediated diseases.Preclinical studies of the mechanism of action suggest that the therapeutic effects afforded by MSC transplantation are short-lived and related to dynamic, paracrine interactions between MSCs and host cells.Clinical trials of MSCs thus far have shown no adverse reactions to allogeneic versus autologous MSC transplants. Clinical studies showed that umbilical cord derived MSC is immunologically stable and not toxic.

This study is to evaluate the safety and the tolerability of UC-MSC (Human Umbilical Cord-Derived Mesenchymal Stem Cell).This study is also to investigate the efficacy of this treatment in patients with Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Men and women who are age in the range of 50 to 85
* All women: go into menopause
* Probable Alzheimer's disease as determined by NINCDS-ADRDA criteria
* MMSE score between 3 and 20, both inclusive
* Voluntarily participating subject who sign the consent form

Exclusion Criteria:

* Subject with cancer
* Subject with positive test for Human Immunodeficiency Virus(HIV)
* Subject who cannot undergo Magnetic Resonance Imaging(MRI), computed tomography(CT) screening
* Subject with psychological diseases (i.e. depression, schizophrenia, bipolar disorder, etc)
* Subject with dementia caused by other than Alzheimer's disease (i.e. infection of central nervous system, Creutzfeld-Jacob disease, severe head trauma, Pick's disease, Huntington's disease, and Parkinson's disease)
* Subject with vascular dementia as determined by the clinical criteria of Design Standards Manual(DSM) IV and the imaging criteria of Erkinjuntii
* Subject with severe white matter hyperintensities (WMH); Severe WMH is defined that length of the deep white matter is 25 mm or longer and length of the periventricular capping/banding is 10 mm or longer.
* Subject who have had stroke in 3 months.
* Subject with severe kidney failure (1.5 mg/dL of serum creatinine or more) Hemoglobin < 9.5 g/dL for men, < 9.0 g/dL for women; Total WBC count < 3000/mm3; Total bilirubin ≥ 3 mg/dL
* Subject who is suspect to have active lung diseases based on check X-ray result
* Subject who have been excluded in the subject selection process for this study before
* A platelet count < 150,000/mm3; Plasma prothrombin time(PT)≥ 1.5; the international normalized ratio (INR) or activated partial thromboplastin time(aPTT)≥ 1.5X control value
* Subject who is determined inappropriate by the investigators

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-03; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse event | 10 weeks from post-administration
  All subjects: Follow-up a year Number of participants with adverse event, number of participants with normal range of vital signs and laboratory examination Indexes of safety evaluation: symptom or sign, laboratory examination, adverse reaction rate

SECONDARY OUTCOMES:
Changes from the baseline in Alzheimer' s Disease Assessment Scale-cognitive subscale(ADAS-Cog) at 10 weeks post-dose | 10 weeks from post-administration
  Changes from the baseline in ADAS-cog, Clinician's Interview-Based Impression of Change(CIBIC), mini-mental state examination（MMSE), CIBIC-plus, Activity of Daily Living Scales(ADL), Neuropsychiatric Inventory(NPI), serum transthyretin, amyloid beta and tau in cerebrospinal fluid, Thl/Th2 cytokines in the peripheral blood.

CONTACTS AND LOCATIONS:
Overall Officials: Hu Chen, M.D., Ph.D., Study Chair — Department of Hematopoietic Stem Cell Transplantation, Affiliated Hospital to Academy of Military Medical Sciences; Bin Zhang, M.D. Ph.D., Study Director — Department of Hematopoietic Stem Cell Transplantation, Affiliated Hospital to Academy of Military Medical Sciences; Dongsheng Fan, M.D., Principal Investigator — Department of Neurology,Peking University Third Hospital
Locations (1):
- Department of Hematopoietic Stem Cell Transplantation, Beijing, China